CLINICAL TRIAL: NCT02874599
Title: Cohort Biomonitoring Study to Evaluate the Biocompatibilty of Resin-based Dental Materials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: S57171
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Materials Testing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients (Experimental): Patients who require multiple dental restorations. Teeth will be restored with commercial restorative composites
  Interventions: Procedure: Dental restoration

INTERVENTIONS:
Procedure: Dental restoration — Damaged teeth will be restored

SUMMARY:
Adult patients who require multiple dental restorations will be included in this study. Urine and saliva samples will be taken for determination of bisphenol A levels at several time points, and for analysis of the estrogenic activity using ERE-CALUX.

Also buccal cells will be taken. Next, DNA extraction will be done with a commercial kit. We will determine global alterations in DNA methylation and DNA hydroxymethylation levels using UPLC-MS/MS.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian, adults,

Exclusion Criteria:

* acute or chronic medical condition, presence of oral inflammatory conditions during the previous 2 weeks, chronic disease requiring intake of drugs, exposure to diagnostic X-rays in the previous 2 months, smoking and consumption of alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-05-02 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Urinary bisphenol A levels | 1 year
Salivary bisphenol A levels | 1 year
%DNA methylation | 6 months
%DNA hydroxymethylation | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- BIOMAT, Department of Oral Health Sciences, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No